CLINICAL TRIAL: NCT02742584
Title: A Randomized Comparative Study Correlating Cough Stress Test With Urodynamics And 24 Hour Pad Test In the Evaluation of Stress Urinary Incontinence
Brief Title: Standardization of Cough Stress Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Henderson, MD, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-11-37
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Stress Urinary Incontinence
Keywords: cough stress test; urodynamics; pad test
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental): Cough Stress Test with a comfortably full bladder.
  Interventions: Procedure: Cough Stress Test
- Group B (Experimental): Cough Stress Test with an empty bladder after straight catheterization.
  Interventions: Procedure: Cough Stress Test
- Group C (Experimental): Cough Stress Test with a bladder infused with 200 cc of saline.
  Interventions: Procedure: Cough Stress Test
- Group D (Experimental): Cough Stress Test with the bladder filled to half functional capacity as determined from the largest voided volume recorded in the patient's voiding diary.
  Interventions: Procedure: Cough Stress Test

INTERVENTIONS:
Procedure: Cough Stress Test — Varying bladder volumes during cough stress test.

SUMMARY:
This is a multicenter, prospective, randomized comparative study in which patients are randomized to one of four different bladder volumes and a Cough Stress Test (CST) is performed in both the standing and sitting positions. The goal is to assess the agreement of each CST method with both urodynamics diagnosis of Stress Urinary Incontinence (SUI) and the 24-hour pad test. The primary outcome is to determine what CST method best correlated with either test in the diagnosis of SUI.

DETAILED DESCRIPTION:
This multicenter, prospective randomized study is approved by the Institutional Review Boards at both the University Hospitals Case Medical Center, Cleveland, OH, USA and MetroHealth Hospital, Cleveland, OH, USA (Identifiers 07-11-37 and FWA00003938, respectively). Adult women who presented to the Female Pelvic Medicine and Reconstructive Surgery (FPMRS) outpatient clinics at both the University Hospitals Case Medical Center and MetroHealth Hospital with symptoms of stress, urge, or mixed urinary incontinence and who were recommended by the evaluating staff to undergo urodynamic studies (UDS) are eligible. The staff physician will approach the patient for participation in this study after the standard clinic visit is completed and the initial diagnosis is made. A research coordinator will then explain the study and obtain informed consent if the patient agrees to participate. The patient will then be given instructions for a 24 hour pad test and standardized pads to use. The patient will also be given instructions for a three day voiding diary along with routine instruction regarding the urodynamic procedure. The patient will be asked to perform the 24 hour pad test the day prior to the UDS appointment. The three day voiding diary will be performed during a typical and sequential three day period during the week prior to the UDS. Patients will then asked to bring these items to the UDS appointment.

During the initial appointment with the study coordinator, patients will be randomized to 4 groups (A, B, C, and D). Patients in group A will be scheduled to undergo Cough Stress Test (CST) with a comfortably full bladder. This will be subjectively reported by the patient. Patients in group B will be scheduled to undergo CST with an empty bladder after straight catheterization. Group C patients will be scheduled to undergo CST with a bladder infused with 200 cc of saline. Patients in group D will be scheduled to undergo CST with the bladder filled to half functional capacity as determined from the largest voided volume recorded in the patient's voiding diary. CST will be performed in the standing and sitting position for each patient in each of the above groups. The sequence of performing the standing and sitting CST will be randomly assigned for each patient.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of urinary incontinence as a chief complaint or as the reason for scheduling the clinic visit, and who were to be scheduled to undergo urodynamic (UDS) testing after initial evaluation by their physician

Exclusion Criteria:

* pelvic organ prolapse beyond stage 1 Pelvic Organ Prolapse- Quantification (POP-Q) as diagnosed by the examining physician
* any other clinical diagnosis other than urinary incontinence who undergo UDS testing ( e.g. interstitial cystitis, overactive bladder dry, bladder outlet obstruction)
* were taking alpha agonists or anticholinergic medications within 2 weeks of the testing
* had an elevated Post Void Residual (PVR) >50cc
* any physical or mental disability that would either not allow participation or impede the ability to give fully informed consent
* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Correlation of cough stress test with urodynamics | 30 minutes
  To define how different accepted cough stress test methods correlated with urodynamics in the evaluation of stress urinary incontinence.

SECONDARY OUTCOMES:
24hour pad weight | 24 hours
  To assess if there was any benefit to performing a 24 hour pad test with or without the different cough stress test modalities.

IPD SHARING:
Plan to Share IPD: No